CLINICAL TRIAL: NCT07272915
Title: Performance Evaluation of the Fujifilm Wako Beta-D-glucan Technique and the Number of Determinations in the Diagnosis of Major Invasive Fungal Infections (IFI)
Brief Title: Performance Evaluation of the Fujifilm Wako Beta-D-glucan Technique in the Diagnosis of Major Invasive Fungal Infections (IFI)
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Anne DEBOURGOGNE, PU-PH, Central Hospital, Nancy, France
Other Study IDs: 2024PI143
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Candidemia; Aspergillosis Invasive; Pneumocystosis; Pneumonia (Etiology); IFI
Keywords: Patients with IFI risks
MeSH Terms: conditions — Candidemia; Pneumonia, Pneumocystis; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Beta-1,3/1,6-D-Glucan — BDG test Fujifilm Wako

SUMMARY:
Invasive fungal infections (IFI) are a major concern for immunocompromised or vulnerable patients. Associated mortality is significant and depends on the timeliness of diagnostic and therapeutic management. Consequently, biomarkers play a key role in therapeutic strategies compared to conventional phenotypic techniques, due to their shorter turnaround time. Beta-D-glucan (BDG) is a pan-fungal serum marker that enables the detection of invasive fungal infections (primarily candidiasis, aspergillosis, and pneumocystosis). This marker was initially introduced by CapeCod, and most studies are based on this test. More recently, the Wako test has been proposed and implemented in our center.

Our study aims to report our experience using the Wako test for BDG measurement, focusing on true and false positives.

The objective is to estimate the test performance, within the patient population, and the percentage of confirmed IFI diagnoses when at least two positive Wako test results are observed in the same patient within a consecutive 15-day period.

ELIGIBILITY:
Inclusion Criteria:

* BDG test in CHRU Nancy

Exclusion Criteria:

* other hospitals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at risk of IFI undergoing one or more BDG measurements performed at CHRU Nancy.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
BDG level | day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France